CLINICAL TRIAL: NCT03275415
Title: Routine Administration of Surfactant/Budesonide to Prevent BPD in VLBW With RDS-A Double Blind Study
Brief Title: Intratracheal Budesonide/Surfactant Prevents BPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Medical University (Other)
Collaborators: Taipei Medical University Hospital (Other); National Taiwan University Hospital (Other); Taipei Veterans General Hospital, Taiwan (Other Government); Mackay Memorial Hospital (Other); Chang Gung Memorial Hospital (Other); China Medical University Hospital (Other); Seventh Medical Center of PLA General Hospital (Other); Guangzhou Women and Children's Medical Center (Other); Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: N201705026
Record Dates: First submitted 2017-09-05; First posted 2017-09-07 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2022-06

CONDITIONS: Respiratory Distress Syndrome; Bronchopulmonary Dysplasia
Keywords: BPD; surfactant; budesonide; respiratory distress syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome; Bronchopulmonary Dysplasia | interventions — Budesonide; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This is a double blind randomized trial. The infants will be randomly assigned into 2 groups: Control (C) (curosurf + saline) and Intervention (I) (curosurf+ budesonide).
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double blind randomized trial. The infants will be randomly assigned into 2 groups: Control (C) (curosurf + saline) and Intervention (I) (curosurf+ budesonide).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Active Comparator): Curosurf + budesonide
  Interventions: Drug: budesonide
- Placebo (Placebo Comparator): Curosurf + saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: budesonide — Intra-tracheal instillation of a combination of budesonide/surfactant in preterm infants with RDS to prevent BPD
  Other Names: pulmicort
  Arms: Experimental
Drug: Saline — Intra-tracheal instillation of a combination of saline/surfactant in preterm infants with RDS to prevent BPD
  Other Names: sodium chloride
  Arms: Placebo

SUMMARY:
A double-blind study includes: 1) birth Wt 500-1499 gm, 2) respiratory distress shortly after birth and requires resuscitation 3) failure to NCPAP within 4 hrs after birth, defined as: a) FIO2 ≥ 0.30, pressure > 5cmH2O b) severe retraction c) apnea d) PCO2 ≥ 60 mmHg. Exclusion criteria: 1) lethal cardiopulmonary status 2) severe congenital anomalies.

Given the COVID19 pandemics, the recruitment became difficult. Under the consideration of scientific and practical consideration, we therefore determine to have a sample of 300, (150 in each group), fulfill the criteria of type I error 0.05, type II error 0.10, power 90% and with an expectation of 30 % improvement of primary outcome (from 60 % in control group to 40 % in the intervention group as original presumed).Appropriate amount of placebo will be used as it does not affect the biophysical property of curosurf (PAS abstract 2017 San Francisco). Primary outcome of study is death or BPD defined by NICHD criteria. Follow up study of neuromotor and cognitive function and pulmonary states will be done at 1-2 years of corrected age.

DETAILED DESCRIPTION:
A double-blind study will be conducted in 7 tertiary centers. Inclusion criteria are: 1) birth Wt 500-1499 gm, 2) respiratory distress shortly after birth and requires resuscitation 3) failure to NCPAP within 4 hrs after birth, defined as: a) FIO2 ≥ 0.30, pressure > 5cmH2O b) severe retraction c) apnea d) PCO2 ≥ 60 mmHg. Exclusion criteria: 1) lethal cardiopulmonary status 2) severe congenital anomalies.

The initial sample size was determined based on the expectation of 30% improvement of the primary outcome (BPD/death) in the intervention group (Curosurf + budesonide) (40%), as compared to control group (Curosurf +saline placebo) (60%), specifying a type I error of 0.05 and type II error 0.20. The total number needed was 240 (120 in each group). The study was started in June 2019 before the pandemic of COVID19 and the study went on smoothly in 2019. Because of the smooth enrollment of the patients in 2019, we decided to increase the ability of the study for detecting the intervention effect through increasing the power from 80 % to 90 % (type II error from 0.2 to 0.1 and type I error decreased from 0.05 to 0.02). The total sample size required was estimated to be 350 (170 in each group). Given the COVID19 pandemics, the recruitment became difficult. Under the consideration of scientific and practical consideration, we therefore determine to have a sample of 300, (150 in each group), fulfill the criteria of type I error 0.05, type II error 0.10, power 90% and with an expectation of 30 % improvement of primary outcome (from 60 % in control group to 40 % in the intervention group as original presumed). The changes in sample size had been approved by independent monitoring committee. We expect that the study will be completed in September 2022.

The sample will be stratified based on birth weight (500-749 grams, 750-999 grams and 1000-1499 grams), the presence of clinical chorioamnionitis or not, and site of study.

ELIGIBILITY:
Inclusion Criteria:

* 1) birth Wt 500-1499 gm, 2) respiratory distress shortly after birth and requires resuscitation, 3) failure to NCPAP within 4 hrs after birth, defined as: a) FIO2 ≥ 0.30, pressure > 5 cmH2O b) severe retraction c) apnea d) PCO2 ≥ 60 mmHg.

Exclusion Criteria:

* 1) lethal cardiopulmonary status, 2) severe congenital anomalies.

Ages: 30 Minutes to 4 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 310 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
incidence of death or BPD | 6 months
  Primary outcome of study is death or BPD defined by NICHD criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Tsu F Yeh, M.D., Ph.D., Principal Investigator — Maternal Child Health Research Center, Taipei Medical University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yeh TF, Chen CM, Wu SY, Husan Z, Li TC, Hsieh WS, Tsai CH, Lin HC. Intratracheal Administration of Budesonide/Surfactant to Prevent Bronchopulmonary Dysplasia. Am J Respir Crit Care Med. 2016 Jan 1;193(1):86-95. doi: 10.1164/rccm.201505-0861OC. PMID 26351971
- [Result] Yeh TF, Lin HC, Chang CH, Wu TS, Su BH, Li TC, Pyati S, Tsai CH. Early intratracheal instillation of budesonide using surfactant as a vehicle to prevent chronic lung disease in preterm infants: a pilot study. Pediatrics. 2008 May;121(5):e1310-8. doi: 10.1542/peds.2007-1973. Epub 2008 Apr 21. PMID 18426851
- [Result] Kuo HT, Lin HC, Tsai CH, Chouc IC, Yeh TF. A follow-up study of preterm infants given budesonide using surfactant as a vehicle to prevent chronic lung disease in preterm infants. J Pediatr. 2010 Apr;156(4):537-41. doi: 10.1016/j.jpeds.2009.10.049. Epub 2010 Feb 6. PMID 20138301